CLINICAL TRIAL: NCT04710251
Title: Effectiveness of Using the Speedometer During Colonoscopy: a Prospective, Comparative Trial
Brief Title: Effectiveness of Using the Speedometer During Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Norwegian Department of Health and Social Affairs (Other Government)
Collaborators: Beth Israel Deaconess Medical Center (Other); Oslo University Hospital (Other); University of Oslo (Other); Showa University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2020P001156
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Colonic Polyp; Colonic Adenoma; Adenoma Colon
Keywords: Colonoscopy; Adenoma detection rate; Withdrawal time; Artificial Intelligence
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colonoscopy with the speedometer (Active Comparator)
  Interventions: Device: Speedometer
- Colonoscopy without the speedometer (No Intervention)

INTERVENTIONS:
Device: Speedometer — We will measure and monitor the withdrawal time of colonoscopy with a speedometer.
  Arms: Colonoscopy with the speedometer

SUMMARY:
PURPOSE OF PROTOCOL

Objective:

To evaluate if the speedometer based on the real-time image analysis can help endoscopists increase their withdrawal time, which is defined as time spent examining the colon during withdrawal of the colonoscope, during colonoscopy.

Hypothesis:

The trial hypothesis is that use of the speedometer during colonoscopy will increase the average withdrawal time, which is defined as time spent examining the colon during withdrawal of the colonoscope, by 1.6 minutes, possibly increasing the performance of the participating endoscopists. Our objective is to clarify the clinical benefits of this digital tool in colonoscopy.

Endpoint: Withdrawal time difference between colonoscopies done without the speedometer (control period) and colonoscopies done with the speedometer (intervention period).

ELIGIBILITY:
Inclusion Criteria:

* Both women and men aged 18 years or older undergoing colonoscopy for any indication at Beth Israel Deaconess Medical Center (BIDMC), Boston, USA.

Exclusion Criteria:

* Known colorectal cancer, hereditary colorectal polyposis, inflammatory bowel disease, or past history of colectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Withdrawal time | Through study completion, an average of 1 year
  Withdrawal time difference between colonoscopies done without the speedometer (control period) and colonoscopies done with the speedometer (intervention period).

SECONDARY OUTCOMES:
Adenoma detection rate (ADR) | Through study completion, an average of 1 year
  Adenoma detection rate (ADR) of the participating endoscopists during the control period and the intervention period.
Quality of colonoscopy | Through study completion, an average of 1 year
  Proportion of colonoscopies with withdrawal time ≥ 6 minutes.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barua I, Misawa M, Glissen Brown JR, Walradt T, Kudo SE, Sheth SG, Nee J, Iturrino J, Mukherjee R, Cheney CP, Sawhney MS, Pleskow DK, Mori K, Loberg M, Kalager M, Wieszczy P, Bretthauer M, Berzin TM, Mori Y. Speedometer for withdrawal time monitoring during colonoscopy: a clinical implementation trial. Scand J Gastroenterol. 2023 Jun;58(6):664-670. doi: 10.1080/00365521.2022.2154616. Epub 2022 Dec 15. PMID 36519564